CLINICAL TRIAL: NCT05858008
Title: Feasibility of Implementing Time-restricted Eating in Women With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Pendergast (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Julie Pendergast, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 81627; 3R01DK124774-03S1 (NIH)
Record Dates: First submitted 2023-05-04; First posted 2023-05-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time-restricted eating (Experimental): Participants will have baseline and post-study data collected, including activity/sleep data, metabolic parameters (fasting labs and anthropometric measurements), and cognitive testing. In addition, food timing will be collected throughout the study. Subjects will be educated about the potential health benefits of time-restricted eating and will self-select a 10-hr window, during which all daily calories will be consumed for 8 weeks.
  Interventions: Behavioral: Time-restricted eating

INTERVENTIONS:
Behavioral: Time-restricted eating — Subjects will be educated about the health benefits of time-restricted eating. Each subject will self-select a 10-hour (10hr +/- 1 hr) window aligned with their active phase during which they will consume all daily calories. Subjects will text the time of their first and last daily calories for the duration of the study.

SUMMARY:
This study will investigate the feasibility of implementing a time-restricted eating intervention in females with mild cognitive impairment. Targeted therapeutic interventions that improve cognitive impairment and delay onset of ADRD are particularly important for females, who have twice the lifetime risk of developing AD, compared to males.

DETAILED DESCRIPTION:
This study will investigate the feasibility of implementing a time-restricted eating (TRE) intervention in females with mild cognitive impairment. Data will be collected for 10 weeks. Baseline food timing, activity/sleep, metabolic health (fasting labs and anthropometric measures), and cognitive testing will be collected in the first two weeks. Subjects will then be invited to enroll in a TRE intervention for 8 weeks. Subjects will be educated about the potential health benefits of TRE, and then each subject will self-select a 10-hr window and consume all daily calories during this time frame. Subjects will text the time of their first and last daily calories for the duration of the study. At the end of the 8-week TRE intervention, metabolic, anthropometric, activity/sleep, and cognitive measurements will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal Women
* Age 45-95
* Diagnosis of mild cognitive impairment

Exclusion Criteria:

* Individuals prone to hypoglycemia
* Liver disease
* Taking medications that affect eating behaviors
* Alcohol consumption of >2 drinks per day
* Significant circadian disruption
* Having care-taking responsibilities that significantly affect sleep
* Shift work or irregular lifestyle
* Diagnosed clinical eating disorder
* Participating in a formal weight loss program

Ages: 45 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants adhering to TRE protocol | From enrollment to study completion up to approximately 8 weeks
  The times of first and last meals will be collected from participants with an SMS texting system. Adherence defined as minimum 10 hour (+/- 1hr) TRE window 5 days per week.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Pendergast, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No